CLINICAL TRIAL: NCT00812851
Title: Randomized Placebo-Controlled Crossover Trial With THC (Delta 9-Tetrahydrocannabinol) for the Treatment of Cramps in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: ALS Association (Other)
Responsible Party: PD Dr. Markus Weber, Neuromuscular Diseases Unit, Kantonsspital St.Gallen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THC SG
Record Dates: First submitted 2008-11-21; First posted 2008-12-22 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2008-11

CONDITIONS: Cramps; Amyotrophic Lateral Sclerosis
Keywords: ALS; cramps; THC; Dronabinol
MeSH Terms: conditions — Muscle Cramp; Amyotrophic Lateral Sclerosis | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dronabinol

SUMMARY:
Many patients with ALS experience cramps during the course of the disease. Frequently, cramps occur as the first symptom of the disease, months before the patients notice weakness and wasting. Cramp severity varies from mild, without affecting daily activities and sleep, to disabling, where almost any voluntary muscle activity induces long standing, severely painful cramping. ALS patients who smoke herbal cannabis (marijuana) or drink hemp tea report lessening of cramps and fasciculations. Although, various medications, such as magnesium, quinine sulfate, lioresal, dantrolene, clonazepam, diphenylhydantoin and gabapentin are used for the treatment of cramps in ALS so far, no medication has been of proven benefit. However, a recent pilot study with THC in ALS showed symptomatic effects in "spasms", fasciculations, insomnia and appetite. The aim of the proposed study is to determine the tolerability, safety and efficacy of THC in the treatment of cramps in ALS. The hypothesis is that THC will lessen cramps in ALS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age and have full legal capacity
* Patients must voluntarily give written informed consent
* Patients diagnosed with possible, probable laboratory supported, probable or definite ALS according to the revised El Escorial criteria (Brooks 2000)
* Patients must score severity of cramps on the VAS 5 or more
* Patients must be able to communicate and report adverse events by phone
* Patients must have laboratory parameters within the following limits: Creatinine, Bilirubin,Transaminases less than 3x upper limit of normal
* Patients may take any medication for the treatment of ALS (ALS -specific and -symptomatic) but may not change this medication during the study period
* Patients must not have cannabis or cannabinoids for at least one month prior to the study and agree not to use it at all during the study. They have to have a negative urinary test for cannabinoids at baseline
* Pre-menopausal females must provide negative pregnancy test within fourteen days before beginning of study participation and have to apply adequate (barrier) birth-control methods
* Patients must agree not to drive a vehicle or use dangerous machines during the entire study period

Exclusion Criteria:

* Patients who are not willing or able to sign the consent form. Doubt of investigator concerning compliance of the patient
* Patients who have a history of failure to respond to, or had significant adverse effects from or hypersensitivity to THC or any cannabinoid
* Patients who have significant concomitant illness(-es), or acute, uncontrolled infections, which might make evaluation of treatment and side effects difficult
* Patients with a history of significant psychiatric disorder, explicitly of schizophrenia
* Patients who are current drug abusers, including alcohol abusers
* Patients with severe coronary artery disease or hemodynamically relevant ECG-documented arrhythmia
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
severity of cramps | 2 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland